CLINICAL TRIAL: NCT04412824
Title: Multimodal Neuroimaging of Alcohol Cues, Cortisol Response, and Compulsive Motivation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sara K Blaine, Assistant Professsor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-263 MR 1907; R00AA025401 (NIH)
Record Dates: First submitted 2020-05-24; First posted 2020-06-02 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Catheters, Indwelling; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Beverage Cues (Active Comparator): Participants will complete an MRI with alcohol beverage visual cues and oral alcohol session.
  Interventions: Drug: Intravenous blood draw
- Non-Alcoholic Beverage Cues (Placebo Comparator): Participants will complete an MRI with non-alcoholic beverage cues and oral alcohol session.
  Interventions: Drug: Intravenous blood draw

INTERVENTIONS:
Drug: Intravenous blood draw — In addition to the oral delivery, an IV line will be placed for the purpose of drawing blood during the MRI session
  Other Names: Indwelling catheter for blood draws

SUMMARY:
This study proposes to examine both the peripheral and central nervous system responses when light social drinkers and binge/heavy social drinkers are exposed to visual ethanol cues, followed by oral ethanol. The findings will provide a greater understanding of the brain mechanisms (cerebral blood flow and functional connectivity) underlying the association between stress, cortisol release, alcohol craving, and alcohol stimulant and sedative effects. This knowledge could be significant in developing new therapies for the treatment of alcoholism.

DETAILED DESCRIPTION:
Results from the 2014 National Survey on Drug Use and Health show that 26% of adults in the US engaged in binge drinking in the past month (SAMHSA 2014). Why some people "mature out" of this behavior while others persist may be due to one's physiological response to binge drinking. No previous study has assessed whether disrupted cortisol and neural network responses to alcohol cues may drive the compulsive alcohol consumption seen in binge drinking individuals who do not yet have an AUD.

The investigator will recruit beer drinking, non-smoking men and women ages 21-45 (N=80, equal gender) who are either moderate drinkers or binge/heavy drinkers for two neuroimaging and neuroendocrine assessments to determine if their "real world" drinking behavior, in a prospective one month follow up, can be predicted based upon the cortisol and neural network responses to alcohol cues (with a placebo control, counter-balanced and randomized). Finally, the influence of genetic variation in the FK506-binding protein 5 (FKBP5) gene, which regulates cortisol activity, on the cortisol and neural network responses to alcohol cues will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Binge/Heavy Social Drinkers (HSD): has never met DSM-IV criteria for alcohol or substance dependence; regular alcohol use over the past year of at least 10 drinks per week, including at lease one occasion per week consuming >4 drinks (males) or >3 drinks (females).
* Able to read and write English.
* Light Social Drinkers (LSD): has never met DSM-IV criteria for alcohol or substance dependence; regular alcohol use over the past year of 1-3 drinks per occasion, 1-3 times weekly, with no more than one occasion per month of drinking >4 drinks (male) or >3 drinks (females) (King et al., 2002).
* Do not meet criteria for any Axis I DSM-IV psychiatric diagnoses except for individuals with a past diagnosis of Post-Traumatic Stress Disorder, Major Depressive Disorder, or Obsessive Compulsive Disorder
* Provide negative urine toxicology screens during initial appointments and at admission for IV/fMRI sessions.
* Body Mass Index between 20-35.
* No current or former nicotine dependence.

Exclusion Criteria:

* Meet current criteria for dependence on any psychoactive substance, excluding caffeine.
* Current or past history of alcohol dependence or abuse.
* Any current use of opiates or past history of opiate abuse/dependence.
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or antabuse.
* Any psychotic disorder or current psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders.
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, liver, thyroid pathology; subjects on medications for any medical condition will be excluded.
* Peri and post-menopausal women, and those with hysterectomies.
* Pregnant and lactating women will be excluded.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Neural Blood Flow | During the Procedure: measurements taken at 10, 20, 30 and 45 minutes during the procedure.
  Blood flow is measured in ml/100 grams/minute. The interpretation is that blood flow to that area indicates that region of the brain is responding to the visual alcohol or non-alcoholic beverage cues. Change in blood flow will be calculated as the change (and slope) of measurements taken at 10, 20, 30 and 45 minutes during the procedure.
Change in Cortisol | Before Procedure to 125 minutes after the procedure.
  The units for cortisol are micrograms/deciliter and the interpretation is that amount has been released into the blood stream from the HPA axis in response to alcohol or alcohol cues. Change in Cortisol will be calculated by taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.
Drinking Behavior in daily experience outside of laboratory | Day after Procedure to 30 days after procedure.
  A smartphone app will be used to collect 4 surveys a day for 30 days after completion of both arms. Multilevel modeling will be used to analyze patterns of drinking over time.
Amount of Alcohol Consumed | Immediately after the procedure.
  After exposure to alcoholic beverage and non-alcoholic beverage visual cues, quantity of alcohol consumed in a free choice test will be measured in milliliters.

SECONDARY OUTCOMES:
Changes in Alcohol Urges (AUQ) | Before Procedure to 125 minutes after the procedure.
  The urge to consume alcohol will be measured using the Alcohol Urge Questionnaire (AUQ). The AUQ consists of 8 questions 8-56 total point distribution. The greater the total points, the greater the measured urge to consume alcohol. The change in alcohol urge will be assessed with the taking the change (and slopes) of measurements at 45, 30 and 5 minutes prior to procedure and comparing it to measurements taken at 65, 95, 110, 125 minutes following the procedure.
Stress levels in daily experience outside of laboratory | Post follow-up procedure (30 days)
  A smartphone app will be used to collect 4 surveys a day for 30 days after completion of both arms. Multilevel modeling will be used to analyze subjective experience of stress over time.
Genetic Risk Factors (Single Nucleotide Polymorphisms; SNPs) Association with Cerebral Blood Flow, Craving, and Real world drinking and stress | Post follow up procedure (within 2 years after procedure)
  One sample of whole blood will be obtained and analyzed for genomic associations with other outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Blaine, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University MRI Center, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
HIPAA requirements prohibit sharing of individual data. De-identified group data will be available.

REFERENCES:
- [Derived] Blaine SK, Ridner CM, Campbell BR, Crone L, Claus ED, Wilson JR, West SN, McClanahan AJ, Siddiq AS, Layman IMP, Macatee R, Ansell EB, Robinson JL, Beck DT. IL-6, but not TNF-alpha, response to alcohol cues and acute consumption associated with neural cue reactivity, craving, and future drinking in binge drinkers. Brain Behav Immun Health. 2023 Jun 11;31:100645. doi: 10.1016/j.bbih.2023.100645. eCollection 2023 Aug. PMID 37484196